CLINICAL TRIAL: NCT06285565
Title: A Nurse-led Coaching Programme With Telemonitoring in Heart Failure: Protocol for a Randomized Controlled Feasibility Study
Brief Title: A Nurse-led Coaching Programme With Telemonitoring in Heart Failure
Acronym: INTERCOACH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alberto Dal Molin (Other)
Collaborators: Azienda Ospedaliero Universitaria Maggiore della Carita (Other)
Responsible Party: Sponsor-Investigator, Alberto Dal Molin, Associate Professor, Università degli Studi del Piemonte Orientale Amedeo Avogadro
Organization: Università degli Studi del Piemonte Orientale Amedeo Avogadro (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CE390/2023
Record Dates: First submitted 2024-02-06; First posted 2024-02-29 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Heart Failure; Telemonitoring; Hospitalizations; Feasibility; Mentoring
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: A parallel, open-label randomized controlled feasibility study
Who Masked: Outcomes Assessor
Masking Description: The assessors will collect clinical outcomes by telephone and will be blinded to the group assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nurse-led supported group (Experimental): A supportive program consisting of the following elements will be provided:
  1. Pre-discharge educational meeting. After the patient is deemed stable, an in-hospital educational intervention will be provided by a trained nurse not involved in the clinical pathway. Key topics of self-care management recognized by the European Society of Cardiology will be discussed.
  2. Telephone nurse-led coaching sessions. In this phase, patients will be encouraged to focus on their values and progress towards their goals. The intervention will be customized based on the objectives identified during the initial meeting. The scheduled sessions will occur weekly during the first months and then transition to twice a month thereafter.
  3. Patients will receive education on measuring weight, blood pressure, heart rate, and oxygen saturation at rest, every morning before breakfast. All participants will be provided with a telemonitoring system that transmits data to a web platform via Bluetooth.
  Interventions: Combination Product: Nurse-led telephone coaching intervention with home telemonitoring of vital signs
- Controlled group (No Intervention): The controlled group will receive usual care

INTERVENTIONS:
Combination Product: Nurse-led telephone coaching intervention with home telemonitoring of vital signs — In addition to standard care, the intervention group will receive a nurse-led supportive programme that involves a pre-discharge educational meeting and 6-month telephone coaching sessions. Patient's caregivers will also be invited to participate. After discharge, patients will be asked to measure their vital signs, daily. In case of alteration, the nurse will ascertain the presence of congestion symptoms and decide to reinforce the recommendations for self-management, request a specialist medical consultant, or refer to the emergency services
  Arms: Nurse-led supported group

SUMMARY:
The goal of this pilot interventional study is to assess the feasibility and acceptability of a supportive intervention for patients affected by heart failure. The main questions it aims to answer are:

* Are implementation strategies effective in facilitating participant fidelity?
* What factors contribute to patients' satisfaction with the designed intervention, and how can these be optimized for improved patient experience and adherence?
* Are the methods and tools established the most appropriate to ensure the completeness of the data collection?

Participants will follow a combined intervention consisting of:

1. pre-discharge educational meeting;
2. telephone nurse-led coaching sessions;
3. home telemonitoring of vital signs.

In the main trial, researchers will compare data from the intervention group with a control group to assess whether it reduces hospitalization rates and improves self-care capabilities

ELIGIBILITY:
Inclusion Criteria:

* aged 65 and over
* hospitalized for cardiac decompensation, regardless of ejection fraction (FE) value (preserved or decreased)
* expected to be discharged home will be considered eligible.

Exclusion Criteria:

* Individuals who lack the cognitive and/or physical capabilities (Mini-COG +) for self-monitoring of vital signs, and without a caregiver available to assist them
* people who receive other medical services

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-09-17 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | 6 months
  the proportion of patients who agreed to participate relative to those who fulfilled the inclusion criteria.
Retention rate | 6 months
  the proportion of patients who complete the study and those who consent to participate
Adherence to the coaching intervention | 4 months.
  the number of coaching phone calls scheduled and actualized
Adherence to telemonitoring program | 4 months.
  the proportion of days during which vital signs were measured and sent by the system relative to the total duration of the intervention
Completeness of data collection | baseline, after 3 and 6 months
  number of returned questionnaires.

SECONDARY OUTCOMES:
90- and 180-day all-cause hospital readmissions | Data collection is planned at 3 and 6 months.
90- and 180-day heart failure-related hospital readmissions | Data collection is planned at 3 and 6 months.
90- and 180-day Emergency Departments visits | Data collection is planned at 3 and 6 months.
90- and 180-day General Practioner visits | Data collection is planned at 3 and 6 months.
90- and 180-day oupatient visits | Data collection is planned at 3 and 6 months.
Self-care capacity (Self-Care of Heart Failure Index ) | Data collection is planned at baseline, 3 and 6 months.
  The self-care capacity of the patient encompasses three dimensions: self-care maintenance, self-care monitoring and symptom perception, and self-care management
Self Care - Self-Efficacy Scale | Data collection is planned at baseline, 3 and 6 months.
  Self-care capacity is mediated by self-efficacy perception, which is the individual's belief in their ability to achieve certain goals as a result of their actions, regardless of the challenges and difficulties they may face. A scale consisting of 10 items using a 5-response Likert scale will be utilized
Quality of life (SF-12 scale) | Data collection is planned at baseline, 3 and 6 months.
  The quality of life is a value that integrates objective indicators (physical health, personal circumstances, social relationships, social and economic influences) and subjective ones (such as how the individual responds to objective conditions) related to various dimensions of life and personal values
Anxiety (Hamilton Anxiety Scale ) | Data collection is planned at baseline, 3 and 6 months.
  The detection of anxiety symptoms (psychological and somatic).
Depression (Geriatric Depression Scale) | Data collection is planned at baseline, 3 and 6 months.
  The detection of depressive symptoms of the elderly
Heart Failure Somatic Perception Scale v.3 (HFSPS) | Data collection is planned at baseline, 3 and 6 months.
  The detecion of somatic symptoms of the disease
Mortality | Data collection is planned at 3 and 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: INES BASSO, Dr, Study Chair — Università degli Studi del Piemonte Orientale Amedeo Avogadro
Locations (2):
- Italy (2):
  - Azienda Ospedaliero-Universitaria maggiore della Carità di Novara, Novara
  - Università del Piemonte Orientale Amedeo Avogadro, Novara

IPD SHARING:
Plan to Share IPD: No